CLINICAL TRIAL: NCT01020292
Title: Nelfinavir and Concurrent Radiation and Temozolomide in Patients With WHO Grade IV Glioma
Brief Title: A Trial of the Protease Inhibitor Nelfinavir and Concurrent Radiation and Temozolomide in Patients With WHO Grade IV Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 01309
Record Dates: First submitted 2009-11-23; First posted 2009-11-24 (Estimated); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Glioma
Keywords: Adult subjects with a diagnosis of Grade IV Glioma
MeSH Terms: conditions — Glioma | interventions — Nelfinavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NFV and Concurrent ChemoRads (Experimental)
  Interventions: Drug: Nelfinavir

INTERVENTIONS:
Drug: Nelfinavir

SUMMARY:
This phase I trial will determine safety, dose-limiting toxicities (DLT) and maximum tolerable dose (MTD) of the protease inhibitor, Nelfinavir (NFV), when given with chemoradiotherapy as post-operative therapy for glioblastoma multiforme (GBM). Oral NFV is a standard therapy for patients with HIV and the safety of 1250 mg BID NFV is well-established. Case studies have also reported that HIV patients have received radiotherapy for cancer, while on 1250 mg BID NFV. This is the first trial of oral NFV and chemoradiotherapy for GBM patients. Although unacceptable toxicity is unlikely, two NFV dose levels (625, and 1250 mg BID) will be evaluated in a cohort escalation design of 3-6 subjects. At the MTD, 19 additional subjects will be enrolled to generate pilot data on radiographic response and to evaluate further toxicity. A maximum of 31 subjects will be enrolled on the trial.

DETAILED DESCRIPTION:
Current therapy for GBM GBM is the most frequent primary malignant brain tumor in adults. Prior to the introduction of temozolomide, the median survival was generally less than one year from the time of diagnosis. Standard therapy had consisted of surgical resection to the extent safely feasible, followed by radiotherapy. Adjuvant carmustine, a nitrosourea drug, was commonly prescribed in the United States. Cooperative-group trials had investigated the addition of various chemotherapeutic regimens to radiotherapy but no randomized phase 3 trial of nitrosourea-based adjuvant chemotherapy had demonstrated a significant survival benefit as compared with radiotherapy alone. A metaanalysis based on randomized trials suggested a small survival benefit of chemotherapy, as compared with Template Version: 7 May 2008 IRB APPLICATION page 1 of 8 radiotherapy alone (a 5 percent increase in survival at two years, from 15 percent to 20 percent). To further improve on these survival rates, the European Organization for Research and Treatment of Cancer (EORTC) Brain Tumor and Radiotherapy Groups, and the National Cancer Institute of Canada (NCIC) Clinical Trials Group completed a randomized, multicenter, phase III trial to compare the alkylating agent temozolomide and radiotherapy with radiotherapy alone in patients with newly diagnosed glioblastoma. [1] A total of 573 patients from 85 centers underwent randomization. At a median follow-up of 28 months, the median survival was 14.6 months with radiotherapy plus temozolomide and 12.1 months with radiotherapy alone. The unadjusted hazard ratio for death in the radiotherapy-plus-temozolomide group was 0.63 (95 percent confidence interval, 0.52 to 0.75; P0.001 by the log-rank test). The two-year survival rate was 26.5 percent with radiotherapy plus temozolomide and 10.4 percent with radiotherapy alone. Concomitant treatment with radiotherapy plus temozolomide resulted in grade 3 or 4 hematologic toxic effects in only 7 percent of patients.

Due to this landmark study, GBM patients who have a good performance status are now typically treated with concurrent radiation and temozolomide followed by adjuvant temozolomide. However, this standard therapy still only results in a median survival of about 14.6 months and a progression-free survival of about 6.9 months. Given these low survival rates, new approaches are needed. The addition of a molecularly-targeted therapy to the standard treatment is an approach that merits further investigation.

GBM, Molecular Markers, and Radiosensitization In GBM, PTEN mutations occur in about a third of patients while EGFR or EGFRvIII (truncated EGFR) amplification occurs in up to 40% of patients. These changes have been shown to correlate with a poor prognosis. Over the past decade EGFR and Ras have been shown to modulate tumor radiosensitivity. EGFR has a number of downstream effectors that include Ras and PI3K. EGFR and Ras-mediated radioresistance is mediated, at least in part by PI3K, and phosphorylated Akt (P-Akt) is a good marker for this effect . We have previously shown in head and neck cancer that P-Akt is a good predictor of clinical response to radiation. We and others have shown that blocking PI3K-Akt pathway enhances radiation response in vitro and in vivo. Radiosensitization occurs in cells in which this pathway is constitutively activated but does not occur in cells (such as normal tissues) in which this pathway is not activated. Inhibition of this pathway, therefore, is a promising approach for radiation sensitization. One difficulty in implementing this therapeutic strategy has been obtaining the means to block this deregulated signaling pathway in patients.

We have found that one class of commonly used drugs, the HIV protease inhibitors (HPIs) interfere with PI3K-Akt signaling. These drugs given in combination with reverse transcriptase inhibitors are the mainstay of the current therapeutic regimens for HIV infected patients. The HPIs are peptidomimetics that inhibit the HIV aspartyl protease, a retroviral enzyme that cleaves the viral gag-pol polyprotein and is necessary for the production of infectious viral particles. One prominent side effect of HPI treatment is insulin resistance. Since Akt, plays a key role in the coordinated regulation of growth and metabolism by the insulin/IGFsignaling pathway, we explored the possibility that HPIs might block the PI3K-Akt signaling axis in tumor cells and hence might be used clinically as radiation sensitizers. We tested NFV and found that it inhibited Akt at concentrations that are routinely achieved in patients. NFV also sensitized tumor cells both in vitro and in vivo to radiation. HPIs have been used continuously in patients with well-characterized pharmacokinetics. There are reports of HIV patients on protease inhibitors who have received radiation therapy; no increase in side effects from the radiation have been reported and clinical outcome may be improved.

In summary, there is clearly strong rationale to proceed with a clinical trial of NFV and chemoradiation in GBM:

1. The prognosis in GBM patients is poor with median survival of 14.6 months with best therapy.
2. Preclinical work demonstrates NFV results in down regulation of Akt signaling in cancer cells and results in radiation sensitization.
3. There is a high frequency of Akt activation in GBM, which has been linked to the pathogenesis and maintenance of the tumor.
4. NFV has been shown to be distributed brain tissue while on therapy and is likely to have increased brain penetrance during fractionated radiotherapy when disruption of the blood-brain-barrier may occur.
5. NFV has not been shown to sensitize normal tissues to radiation.
6. NFV has been safely administered to HIV+ patients over the last decade with minimal side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients > 18 years old.
2. Newly diagnosed and histologically confirmed supratentorial WHO Grade IV astrocytoma status-post maximally achievable resection.
3. ECOG performance status 0-2.
4. Absolute Neutrophil Count ≥ 1500 per mm3
5. Platelet count ≥ 100,000 per mm3
6. Serum creatinine < 1.5 times the upper limit of normal
7. Serum AST or ALT < 2 times the upper limit of normal
8. Serum bilirubin < 1.5 mg/dl
9. Patients who were receiving corticosteroids have to receive a stable or decreasing dose for at least 14 days before randomization.
10. No prior cranial radiotherapy will be permitted.
11. No known HIV infection.
12. The effects of NFV on the developing human fetus have been studied in HIV positive women.

    We do not, however, know the risks along with radiation. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
13. Patients must sign an informed consent document that indicates they are aware of the investigative nature of the treatment in this protocol as well as the potential risks and benefits.

Exclusion Criteria:

1. Prior cranial radiotherapy.
2. Patients may not be receiving or have received any other investigational agents during/or within 1 month prior to treatment with NFV.
3. Pregnant or lactating women.
4. Patients receiving the following drugs that are contraindicated with NFV will be excluded: antiarrhythmics (amiodarone, quinidine), antimycobacterial (rifampin), ergot derivatives (dihydroergotamine, ergonovine, ergotamine, methylergonovine), herbal products (St. John's wort), HMG-CoA reductase inhibitors (lovastatin, simvastatin), neuroleptic (pimozide), proton pump inhibitors, sedatives/hypnotics (midazolam, triazolam).
5. Patients receiving the following drugs will be clinically evaluated as to whether dosage/medication can be changed to permit patient on study: anti-convulsants (carbamazepine, phenobarbital, phenytoin), anti-mycobacterial (rifabutin), PDE5 inhibitors (sildenafil, vardenafil, tadalafil), HMG-CoA reductase inhibitor (atorvastatin, rosuvastatin), immunosuppressants (cyclosporine, tacrolimus, sirolimus), narcotic analgesic (methadone), oral contraceptive (ethinyl estradiol), macrolide antibiotic (azithromycin), antidepressant (trazadone).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
To determine the safety, dose-limiting toxicities, and maximally tolerated dose of NFV concurrently with radiation and temozolomide. | One year

SECONDARY OUTCOMES:
To determine the progression free survival (PFS) and overall survival (OS) with an exploratory analysis to compare the observed median value obtained in this study to the historical median values of 6.9 months and 14.6 months respectively. | Two years

CONTACTS AND LOCATIONS:
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States